CLINICAL TRIAL: NCT01162668
Title: Assessment of Outcomes Following Bariatric Surgery for Mississippi State Employees
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Katie McClendon, Clinical Assistant Professor, University of Mississippi Medical Center
Other Study IDs: 41165
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: bariatric surgery; obesity; outcomes
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: to assess the health and economic outcomes (weight lost, change in control of chronic diseases such as diabetes, quality of life, work productivity, health care cost, etc) associated with bariatric (weight-loss) surgery for 200 severely obese patients who undergo bariatric surgery as part of the Mississippi State Employees' Life and Health Insurance Plan's Obesity Treatment Program (OTP).

2. Patient Characteristics: Inclusion criteria: Eligible bariatric surgical candidates who are enrolled in the OTP (100 patients per year for 2 years). The Plan's criteria includes, but is not limited to 1) enrollment in the plan for at least 12 consecutive months prior to September 1, 2009; 2) completion of the HealthQuotient health risk assessment through the Plan's wellness and health promotion program; 3) a Body Mass Index (BMI) of >40 kg/m2, or a BMI >35 kg/m2 with two or more co-morbidities such as diabetes, hypertension, sleep apnea or asthma; 4) two or more physician-supervised weight loss attempts within the last 24 months; 5) age 18 years or older; and 6) consent to provide personal and medical information to the Plan. Prior to surgery, each site administers a psychiatric evaluation to ensure the patient is psychologically stable for surgery. Exclusion criteria: any patient who does not meet criteria above or who declines to participate. Surgeries will take place only at Certified Bariatric Surgery Centers of Excellence (COE), of which, there are currently 3 in the state. The 3 COEs exist with 4 outpatient medical offices (1 COE is composed of 2 independent surgeon practices) Patients will be recruited at each site once they are approved by the OTP.

3. Design: prospective, observational, multi-center, longitudinal study of outcomes and resource utilization associated with OTP. Estimates of obesity and comorbidities' impact will be obtained from the outpatient medical office for the COEs. Medical charts, databases and medical/pharmacy claims will be the source of information. Surveys on quality of life, productivity, and patient satisfaction will be administered directly to patients. Database claim information will be obtained in future and is not a part of current IRB application.

4: Procedures: After obtaining informed consent, patients will be administered surveys at baseline, as well as at follow-up visits. Additional data will be obtained via patient charts, databases, and medical/pharmacy claims.

ELIGIBILITY:
Inclusion Criteria:

* Eligible bariatric surgical candidates who are enrolled in the Mississippi SSELHI Plan (100 candidates enrolled per year). The Plan's criteria includes, but is not limited to

  1. enrollment in the plan for at least 12 consecutive months prior to September 1, 2009
  2. completion of the HealthQuotient health risk assessment through the Plan's wellness and health promotion program
  3. a Body Mass Index (BMI) of >40 kg/m2, or a BMI >35 kg/m2 with two or more co-morbidities such as diabetes, hypertension, sleep apnea or asthma
  4. two or more physician-supervised weight loss attempts within the last 24 months
  5. consent to provide personal and medical information to the Plan

Exclusion Criteria:

* Any patient who does not meet criteria above or who declines to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 obese patients with Mississippi State Employee Insurance who undergo bariatric surgery as part of Obesity Treatment Program
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Weight loss | 0, 6, 12, and 24 months
  change in weight from baseline
Body mass index (BMI) | 0, 6, 12, and 24 months
  Change in body mass index (BMI) from baseline

SECONDARY OUTCOMES:
ecomonic outcomes | 0, 6, 12, and 24 months
  costs to the insurance plan were assessed
Systolic blood pressure | 0, 6, 12, and 24 months
  change in systolic blood pressure from baseline
Diastolic blood pressure | 0, 6, 12, and 24 months
  change in diastolic blood pressure from baseline
Medication use | 0, 6, 12, and 24 months
  Change in mean number of medications prescribed
quality of life | 0, 6, 12, and 24 months
  Impact of weight on quality of life (IWQOL-lite) questionnaire; tool assesses 5 domains of quality of life: physical function, self-esteem, sexual life, public distress, and work impact
Work productivity | 0, 6, 12, and 24 months
  Work productivity and activity impairment questionnaire: General Health v2.0 (WPAI:GH) assesses work productivity

OTHER OUTCOMES:
Surgery-related adverse events | 24 months
  Any surgery-related adverse events were noted

CONTACTS AND LOCATIONS:
Overall Officials: Katie S McClendon, Pharm.D., Principal Investigator — University of Mississippi Medical Center
Locations (4):
- United States (4):
  - Central Mississippi Medical Center Comprehensive Weight Management Program, Jackson, Mississippi
  - Oxford Bariatric, Oxford, Mississippi
  - Oxford Surgical & Bariatric Clinic,LLC., Oxford, Mississippi
  - South Mississippi Surgical Weight Loss Center, Pascagoula, Mississippi

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-04-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT01162668/Prot_SAP_000.pdf
  • Informed Consent Form (2012-04-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT01162668/ICF_001.pdf